CLINICAL TRIAL: NCT04701749
Title: Study of the Effects of Anticoagulant Interruption Covered by Percutaneous Left Atrial Occlusion in Patients With Chronic Atrial Fibrillation and Radiation Cystitis at Risk of Bleeding
Acronym: HEMOCC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2020 GUY; 2020-A02246-33 (Other: 2020-A02246-33)
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Radiation Cystitis; Non-valvular Atrial Fibrillation
Keywords: radiation cystitis; Hematuria; Left atrial appendage closure or left atrial occlusion (LAO)
MeSH Terms: conditions — Hematuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with atrial closure
  Interventions: Device: Percutaneous left atrial closure
- without atrial occlusion
  Interventions: Other: No Percutaneous left atrial closure

INTERVENTIONS:
Device: Percutaneous left atrial closure — Percutaneous left atrial closure was performed under general anesthesia with angiographic control and transesophageal echocardiography. The procedure takes between 15 and 20 minutes. This begins with a right femoral venipuncture, progression of the guide in the right atrium allowing atrial trans-septal puncture to catheterize the left atrium. A nitinol prosthesis is implanted (Boston Watchman) at the ostium of the left auricle between the left superior pulmonary vein and the circumflex artery. After a tensile test verifying the stability of the prosthesis, the absence of peri-prosthetic leakage is verified by ETO and angiographic control. The patient is monitored 48 hours before discharge to eliminate the appearance of pericardial effusion and prosthetic embolization. Aspirin 75 mg monotherapy is started the same day with stopping anticoagulation.
  Groups: with atrial closure
Other: No Percutaneous left atrial closure — No Percutaneous left atrial closure
  Groups: without atrial occlusion

SUMMARY:
The etiology of the radiation cystitis is a pelvic irradiation generally performed as part of the treatment of prostate cancer. The incidence is 50,000 new cases per year. Approximately 35% of prostate cancer treatment is radiotherapy. The prevalence of haematuric radiation cystitis is 4-5% (about 800 patients).

One of the complications of radiation cystitis is persistent hematuria. There is currently no curative treatment for this hematuria. There are few treatment options with a random probability of improvement of this symptomatology. These haematurias are rarely resolved spontaneously and most of the time involve emergency room management with +/- invasive procedures, sometimes by hospitalisation, always with a significant psychological impact on the patient.

Furthermore, lifetime anticoagulant treatment considerably increases the likelihood of bladder bleeding. This is the case of patients being followed for Atrial Fibrillation Cardiac Arrhythmia (AFCA), which by definition carries a major cardioembolic risk, and who will be of particular interest in this study.

In recent years, cardiologists have developed an alternative to anticoagulants: left atrial appendage closure or left atrial occlusion (LAO) . This procedure consists of inserting a nitinol prosthesis in the left atrium, the site of more than 90% of thrombi formation in non-valvular atrial fibrillation. This minimally invasive procedure lasts about 15 minutes and is performed during a 48-hour hospitalization. Anticoagulants are stopped the day after the setting up procedure. Several studies have shown non-inferiority of atrial closure and anticoagulants to thromboembolic events in non-valvular atrial fibrillation. In addition, LAO allows the permanent discontinuation of anticoagulants, associated with the cessation of anticoagulant bleeding adverse events.

While studies have been conducted on the impact of this technique on patients monitored in cardiology, no studies evaluate the value of LAO in anticoagulated patients with a hematuric radiation cystitis. This tprocedure is already used in routine care for patients followed in urology, and has shown encouraging results, since 8 out of 10 patients saw a significant reduction in the number of haematurias, but it has never yet been scientifically proven to be effective, hence the aim of this study.

The interest of this study will therefore be :

* To evaluate the potential benefit of left atrial appendage closure on the number of episodes of hematuria.
* To evaluate the economic benefit in reducing the number of hospitalizations, surgeries and complications for hematuria as well as the discontinuation of anticoagulants.

As the patient's data must be retrieved regardless of the patient's subsequent management (with or without a cardiac procedure) within the framework of the HEMOCC protocol, it will be proposed to the patient as soon as he or she is consulting for haematuria on radiation cystitis. The patient will be followed for 3 years.

The mainly descriptive analyses will be collected in the form of a register and carried out by a biostatistician from Clermont-Ferrand University Hospital.

DETAILED DESCRIPTION:
Prospective single-centre observational study involving the creation of a data registry of patients with anticoagulation-treated non-valvular atrial fibrillation with hematuria on radiation cystitis.

Patients who present a hematuria on radial bladder associated with anticoagulated atrial fibrillation will be recruited into the protocol by an urologist from Gabriel MONTPIED UHC once they have presented at least one episode of hematuria on radial bladder under anticoagulant treatment in the context of a non-valvular ACFA, and once they have given their agreement to participate in the HEMOCC research protocol.

A research associate will meet the patient to finalize the administrative and practical aspects of inclusion and the collection of retrospective data. Regardless of whether or not left atrial occlusion is performed, the patient's data included in the protocol will be collected.

The urologist will then refer the patient to Pr ESCHALIER's cardiology department for cardiological advice regarding an indication of percutaneous occlusion of the left atrium (running walk).

If LAO is indicated and the patient agrees to the procedure, then the procedure will be scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old benefiting a social security sheme.
* Patient with hematuric radiation bladder associated with a non valvular anticoagulated atrial fibrillation.

Exclusion Criteria:

* All the other hematuria's reasons
* Other reason of anti platelet agent using than atrial fibrillation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with at least one hematuria while on anticoagulant therapy for non-valvular atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants | Baseline (Month 0)
  number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants collected with a data collection form
number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants | Month 3
  number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants collected with a data collection form
number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants | Month 6
  number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants collected with a data collection form
number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants | Month 9
  number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants collected with a data collection form
number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants | Month 12
  number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants collected with a data collection form
number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants | Month 18
  number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants collected with a data collection form
number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants | Month 24
  number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants collected with a data collection form
number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants | Month 30
  number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants collected with a data collection form
number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants | Month 36
  number of episodes of hematuria following atrial occlusion and discontinuation of anticoagulants collected with a data collection form

SECONDARY OUTCOMES:
Number of days hospitalizations for hematuria | Baseline (Month 0)
  assessed by phone contact
Number of days hospitalizations for hematuria | Month 3
  assessed by phone contact
Number of days hospitalizations for hematuria | Month 6
  assessed by phone contact
Number of days hospitalizations for hematuria | Month 9
  assessed by phone contact
Number of days hospitalizations for hematuria | Month 12
  assessed by phone contact
Number of days hospitalizations for hematuria | Month 18
  assessed by phone contact
Number of days hospitalizations for hematuria | Month 24
  assessed by phone contact
Number of days hospitalizations for hematuria | Month 30
  assessed by phone contact
Number of days hospitalizations for hematuria | Month 36
  assessed by phone contact
duration of hematuria episodes | Baseline (Month 0)
  assessed by phone contact
duration of hematuria episodes | Month 3
  assessed by phone contact
duration of hematuria episodes | Month 6
  assessed by phone contact
duration of hematuria episodes | Month 9
  assessed by phone contact
duration of hematuria episodes | Month 12
  assessed by phone contact
duration of hematuria episodes | Month 18
  assessed by phone contact
duration of hematuria episodes | Month 24
  assessed by phone contact
duration of hematuria episodes | Month 30
  assessed by phone contact
duration of hematuria episodes | Month 36
  assessed by phone contact
number of hematuria surveys | Baseline (Month 0)
  assessed by phone contact
number of hematuria surveys | Month 3
  assessed by phone contact
number of hematuria surveys | Month 6
  assessed by phone contact
number of hematuria surveys | Month 9
  assessed by phone contact
number of hematuria surveys | Month 12
  assessed by phone contact
number of hematuria surveys | Month 18
  assessed by phone contact
number of hematuria surveys | Month 24
  assessed by phone contact
number of hematuria surveys | Month 30
  assessed by phone contact
number of hematuria surveys | Month 36
  assessed by phone contact

CONTACTS AND LOCATIONS:
Overall Officials: Laurent GUY, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France